CLINICAL TRIAL: NCT01129024
Title: An Open-label Safety Study of S-888711 in Adult Subjects With Relapsed Persistent or Chronic Immune Thrombocytopenia With or Without Prior Splenectomy
Brief Title: An Open-label Safety Study of Lusutrombopag (S-888711) in Adults With Chronic Immune Thrombocytopenia (ITP)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to cessation of clinical development of S-888711 for chronic ITP based on a business decision by the Sponsor.
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0914M0622
Record Dates: First submitted 2010-05-07; First posted 2010-05-24 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Immune Thrombocytopenia
Keywords: Splenectomy; Low Platelet Count; Thrombopoiesis; Thrombocytopaenia; Idiopathic Thrombocytopenic Purpura; Immune Thrombocytopenia (ITP); Thrombotic Thrombocytopenic Purpura (ITP); Hematologic Disease; Auto-immune Thrombocytopenic Purpura; S-888711; Blood Platelet Disorders; Relapsed Persistent or Chronic ITP; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Purpura, Thrombotic Thrombocytopenic; Hematologic Diseases; Blood Platelet Disorders | interventions — lusutrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lusutrombopag (Experimental): Participants received lusutrombopag 0.5 mg administered orally once a day for up to 3 years or until study termination. The dose was adjusted based on platelet counts. If a subject's platelet count remained < 50,000/μL, the dose could have been increased by 0.25 mg up to a maximum dose of 2.0 mg.
  Interventions: Drug: Lusutrombopag

INTERVENTIONS:
Drug: Lusutrombopag — tablet
  Other Names: MULPLETA®; S-888711

SUMMARY:
The primary objective of this study was to assess the long-term safety of lusutrombopag in the treatment of adults with relapsed persistent or chronic ITP with or without prior splenectomy.

DETAILED DESCRIPTION:
This was an open-label, long-term safety study of lusutrombopag in the treatment of adults with relapsed persistent or chronic ITP with or without prior splenectomy. Patients who participate in this study must have completed the Phase 2 study 0913M0621 (NCT01054443), a double-blind, placebo controlled, parallel group study that evaluated the efficacy and safety lusutrombopag during which they either completed treatment or discontinued treatment due to a platelet count > 400,000/μL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who previously participated in Study 0913M0621 (NCT01054443) and who completed treatment or discontinued treatment due to a platelet count > 400,000/μL and continued to meet all inclusion criteria of the previous study, listed below, including platelet counts < 50,000/μL were eligible for study participation. For the purpose of this study, initial screening visit and all prestudy time period refer to Study 0913M0621.
* A signed and dated written informed consent
* Males and females ≥ 18 years of age
* All subjects must agree to use barrier contraception
* Diagnosis of ITP
* Subjects > 60 years must have had a diagnostic bone marrow aspiration
* Relapsed persistent or chronic ITP status, with or without prior splenectomy
* Subjects receiving steroid therapy must be on a stable dose for at least 2 weeks prior to Screening
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) within 20% of the upper limit of normal (ULN) at Screening
* Subjects receiving stable dosages of cyclosporine A, mycophenolate mofetil, azathioprine, or danazol are allowed

Exclusion Criteria:

* History of clinically important hemorrhagic clotting disorder
* Females who are pregnant, lactating, or taking oral contraceptives
* History of alcohol/drug abuse or dependence within 1 year
* Use of the following drugs or treatment prior to Visit 1 (Day 1):

  * Within 1 week - Rho(D) immune globulin or intravenous immunoglobulin;
  * Within 2 weeks - plasmaphoresis treatment;
  * Within 4 weeks - use of anti-platelet or anti-coagulant drugs;
  * Within 8 weeks - rituximab;
  * Within 12 weeks - alemtuzumab, multi-drug systemic chemotherapy, stem cell therapy;
* History of clinically significant cardiovascular or thromboembolic disease within 26 weeks prior to Initial Screening
* Splenectomy within 4 weeks prior to Initial Screening
* Clinically significant laboratory abnormalities

  * Hemoglobin < 10.0 g/dL for men or women, not clearly related to ITP
  * Absolute neutrophil count < 1000/mm3
  * Abnormal peripheral blood smear with evidence of fibrosis confirmed by bonemarrow biopsy
  * Total bilirubin > 1.5 x upper limit of normal
  * Alanine aminotransferase (ALT) > 1.5 x upper limit of normal
  * Aspartate aminotransferase (AST) > 1.5 x upper limit of normal
  * Creatinine > 1.5 x upper limit of normal
  * Human immunodeficiency virus positive
  * Hepatitis A IgM antibody positive, hepatitis B surface antigen or hepatitis C antibody positive
* Exposure to previous thrombopoietin (TPO) mimetics/agonists (e.g., eltrombopag,romiplostim, E5501 [AKR-501] or LGD-4665) within 4 weeks prior to Initial Screening
* Subjects unresponsive to previous TPO mimetics/agonists (e.g., eltrombopag, romiplostim, E5501 [AKR-501] or LGD-4665)
* Exposure to an investigative medication within 4 weeks prior to the initial Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04-29 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (18):
- United States (18):
  - Investigator, Anaheim, California
  - Investigator, Los Angeles, California
  - Investigator, Washington D.C., District of Columbia
  - Investigator, Boynton Beach, Florida
  - Investigator, Jacksonville, Florida
  - Investigator, Atlanta, Georgia
  - Investigator, Riverdale, Georgia
  - Investigator, Metairie, Louisiana
  - Investigator, Bethesda, Maryland
  - Investigator, Boston, Massachusetts
  - Investigator, Jefferson City, Missouri
  - Investigator, Kansas City, Missouri
  - Investigator, New Brunswick, New Jersey
  - Investigator, New York, New York
  - Investigator, Cleveland, Ohio
  - Investigator, San Antonio, Texas
  - Investigator, Salt Lake City, Utah
  - Investigator, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who previously participated in Study 0913M0621 (NCT01054443) and who completed treatment or discontinued treatment due to a platelet count > 400,000 cells/μL were rolled over into this open-label extension study.
Groups:
- Lusutrombopag: Participants received lusutrombopag 0.5 mg administered orally once a day for up to 3 years or until study termination. The dose was adjusted based on platelet counts.
Period: Overall Study
Arm/Group | Lusutrombopag
Started | 19
Completed | 0
Not Completed | 19
Not completed — Physician Decision | 5
Not completed — Study Terminated by Sponsor | 8
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 3
Not completed — Needed a Platelet Transfusion | 1

BASELINE CHARACTERISTICS:
Population: All enrolled and treated participants
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (20.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18
  Black or African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An AE is defined as any untoward medical occurrence in a subject administered a pharmaceutical product during the course of a clinical investigation, including any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product (IP), whether or not thought to be related to the IP. AEs reported after initial study drug administration were considered treatment-emergent.
  A serious adverse event is defined as any AE that resulted in death, was life-threatening, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect or an important medical event that, based upon medical judgment, may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed above.
  A treatment-related AE is any AE determined by the investigator to be possibly related, probably related, or definitely related to study drug.
Time Frame: From first dose of study drug in the extension study up to 6 weeks after last dose; median (range) time on study treatment was 148 (10-387) days.
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 19
Participants
  Any treatment-emergent adverse event (TEAE) | 19
  Serious TEAEs | 1
  Treatment-related TEAEs | 3
  Treatment-related serious TEAEs | 0
  TEAEs leading to study discontinuation | 2

2. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the percentage of the cumulative time a platelet count was ≥ 50,000 cells/µL during the extension study.
Time Frame: From first dose of study drug in the extension study up to 6 weeks after last dose; median (range) time on treatment was 148 (10 - 387) days.
Population: All enrolled and treated participants
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 19
percentage of days | 0.200 [0.00 to 0.80]

3. Secondary Outcome: Number of Participants With Worst Severity of Bleeding Associated With ITP During the Treatment Period
Description: Bleeding assessments were performed by the Investigator according to the World Health Organization (WHO) criteria bleeding scale:
  Grade 0: no bleeding; Grade 1: petechial bleeding; Grade 2: mild blood loss (clinically significant); Grade 3: gross blood loss, requires transfusion (severe); Grade 4: debilitating blood loss, retinal or cerebral associated with fatality.
  For each participant, the most severe WHO bleeding grade observed during the treatment period is reported.
Time Frame: Bleeding assessments were performed at Weeks 1, 2, 3, 4, 5, and 6, Months 1, 2, 3, 6, 9, and 12, and every 3 months thereafter until end of treatment; median (range) time on treatment was 148 (10-387) days.
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 19
Participants
  Grade 0 | 3
  Grade 1 | 11
  Grade 2 | 5
  Grade 3 | 0
  Grade 4 | 0

4. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count of < 50,000 Cells/μL, Between 50,000 to 400,000 Cells/μL, and ≥ 400,000 Cells/μL
Description: This analysis includes platelet counts measured during the treatment period, including while participants were taking rescue medications.
Time Frame: Platelets were assessed at Weeks 1, 2, 3, 4, 5, and 6, Months 1, 2, 3, 6, 9, and 12, and every 3 months thereafter, until end of treatment; median (range) time on treatment was 148 (10-387) days.
Population: All enrolled and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 19
percentage of participants
  Platelet count < 50,000 cells/μL | 31.6
  Platelet count ≥ 50,000 and < 400 cells/μL | 68.4
  Platelet count ≥ 400,000 cells/μL | 0.0

5. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count of < 50,000 Cells/μL, Between 50,000 to 400,000 Cells/μL, and ≥ 400,000 Cells/μL Without Rescue Medication
Description: This analysis excludes platelet counts measured while the participant was taking rescue medications and during the 4 weeks after rescue medication.
Time Frame: as for outcome 4
Population: All enrolled and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 19
percentage of participants
  Platelet count < 50,000 cells/μL | 42.1
  Platelet count ≥ 50,000 and < 400,000 cells/μL | 57.9
  Platelet count ≥ 400,000 cells/μL | 0.0

6. Secondary Outcome: Change From Baseline in Platelet Counts at the Final Visit
Time Frame: Baseline and the final visit (If a subject had multiple platelet count measurements for the specific dose level due to dose adjustments, the final platelet count was used)
Population: All enrolled and treated participants
Measure: Median (Full Range); unit: cells/μL
Arm/Group | Lusutrombopag
Number analyzed (Participants) | 19
cells/μL
  Baseline | 23000.00 [9000.0 to 40000.0]
  Final visit | 23000.00 [4000.0 to 124000.0]
  Change from Baseline | 3000.00 [-19000.0 to 108500.0]

ADVERSE EVENTS:
Time Frame: From first dose of study drug in the extension study up to 6 weeks after last dose; median (range) time on study treatment was 148 (10-387) days.
Arm/Group | Lusutrombopag
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lusutrombopag (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Suicidal ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lusutrombopag (N=19)
Nasopharyngitis (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Burn infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Mouth haemorrhage (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Salivary gland disorder (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 6
Oedema peripheral (General disorders) | 2
Cyst (General disorders) | 1
Pain (General disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Blood blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Bone marrow reticulin fibrosis (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Affective disorder (Psychiatric disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Mood disorder due to a general medical condition (Psychiatric disorders) | 1
Personality disorder (Psychiatric disorders) | 1
Polysubstance dependence (Psychiatric disorders) | 1
Tachyphrenia (Psychiatric disorders) | 1
Blood potassium decreased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Myodesopsia (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Breast fibrosis (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Breast tenderness (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Balance disorder (Nervous system disorders) | 1
Carotid artery disease (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Haematoma (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Phlebitis superficial (Vascular disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.